CLINICAL TRIAL: NCT02139254
Title: First Trimester Glycosylated Haemoglobin Und Plasma Glucose in Women at High Risk for Gestational Diabetes
Acronym: GDM HbA1c
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 030/13
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; HbA1c; Glucose; First Trimenon
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low risk: Pregnant women with a low risk for metabolic diseases
- High risk: Pregnant women with a high risk for metabolic diseases

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as carbohydrate intolerance with onset or first recognition during pregnancy. If insulin resistance and hyperglycemia are recognized before pregnancy, the term pregestational diabetes (PGD) is used. In the last years, much has been invested to uniformly define worldwide the diagnostic criteria and the management of gestational diabetes. A general screening in a low risk population should be implemented into routine prenatal care. Similarly, pregnant women at high risk for metabolic disorders should be screened in the early pregnancy.

The aim of the following study ist to investigate the role of first trimester glycosylated haemoglobin (HbA1c) of pregnant women with risk factors in developing gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Background

Gestational diabetes mellitus (GDM) is defined as carbohydrate intolerance with onset or first recognition during pregnancy. If insulin resistance and hyperglycemia are recognized before pregnancy, the term pregestational diabetes (PGD) is used. In the last years, much has been invested to uniformly define worldwide the diagnostic criteria and the management of gestational diabetes. Recently, the American Diabetes Association stated that a general screening in a low risk population should be implemented into routine prenatal care. However, there are still controversies on which diagnostic criteria to use. Similarly, screening of pregnant women at high risk for PGD is also a matter of debate. This is an important issue as the prevalence of this group is increasing worldwide. Of interest, the ADA as well as the international expert committee on diabetes published a consensus statement in which the use of HbA1c was supported for the diagnosis of diabetes rather than the measurement of fasting or post-prandial plasma glucose in a non-pregnant population. A value of ≥6.5% (≥48mmol/mol) was proposed as criterion for diagnosis. There is no doubt that the measurement of glycosylated haemoglobin may be of value in particular preconceptional in diabetes type 1. Difference exist in using HbA1c during pregnancy. At the pregnant state, the different red cell turnover and other physiologic changes in pregnancy may interfere with HbA1c. Indeed, mean HBA1c levels in healthy pregnant women are lower than in the non-pregnant women. Moreover, O'Connor et al. showed that first and second trimester HbA1c values are significantly different to a non-pregnant population, whereas no difference was found comparing HbA1c values from the third trimester. Therefore, it has been suggested, that only blood glucose criteria should be used to diagnose or exclude PGD in particular during the first trimester as the data on HBA1c in the first trimester is limited .

Objective

To observe the values of HbA1c obtained from pregnant women in the early pregnancy, the difference between those who develop GDM and those who do not and the comparison of first trimester HBA1c, Plasma Glucose and angiogenesis factors.

Methods

This is an observational prospective cohort study conducted in our Department of Obstetrics. All women are tested for HbA1c at the first antenatal visit during the first trimester. First trimester was defined as up to 12 6/7 weeks of gestation. Between 24 and 28 weeks of gestation the women are screened, as internationally proposed, by a "one-step" standardized 75g oral glucose tolerance test (oGTT). Venous blood samples were collected at 0, 1, and 2h after the glucose load. Women with pre-existing diabetes mellitus or a first trimester HbA1c ≥6.5% are excluded from the study und medical care for pregestational diabetes is provided.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* 8-13 weeks of gestation
* Written informed consent

Exclusion Criteria

* Pregestational diabetes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who receive antenatal care at the Department of Obstetrics in our Hospital and have the first vist between 8. and 12. week of pregnancy. Women with pregestational diabetes are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Number of women with gestational diabetes | Week 28 of pregnancy

SECONDARY OUTCOMES:
Delivery Mode | At delivery, expected to be on average after 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Raio, PD, Principal Investigator — Frauenklinik Inselspital Bern
Locations (1):
- Dep. of Obstetrics and Gynecology, Bern, Switzerland

REFERENCES:
- [Derived] Amylidi-Mohr S, Lang C, Mosimann B, Fiedler GM, Stettler C, Surbek D, Raio L. First-trimester glycosylated hemoglobin (HbA1c) and maternal characteristics in the prediction of gestational diabetes: An observational cohort study. Acta Obstet Gynecol Scand. 2023 Mar;102(3):294-300. doi: 10.1111/aogs.14495. Epub 2022 Dec 16. PMID 36524557